CLINICAL TRIAL: NCT05684523
Title: Feasibility Study on the Use of Redormin® 500 (Ze 91019) on Day-time Cognition and Quality of Life in People With Occasional Sleep Problems
Brief Title: Feasibility Study on the Use of Redormin®500 on Day-time Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max Zeller Soehne AG (Industry)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Ze 91019-04-2022-01
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disorders, Circadian Rhythm; Cognitive Dysfunction
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Cognitive Dysfunction | interventions — Hova

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Redormin® 500 (Experimental): fixed combination of valerian and hops dry extract, 500 mg, once daily for 21 days
  Interventions: Drug: Valerian-Hop Extract
- Placebo (Placebo Comparator): matching placebo, once daily for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valerian-Hop Extract — herbal drug
  Other Names: Redormin® 500
  Arms: Redormin® 500
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, parallel groups, placebo-controlled, baseline/run-in period of 21 days followed by trial period of 21 days, digital phenotyping (sleep, cognitive/psychological parameters and HRV).

The aim of this study is to determine the feasibility of investigating the effects of Redormin® 500 on day-time cognition and to assess psychological parameters (subjective cognitive performance, tiredness, mood, stress level, quality of life, motivation), in people with occasional sleep problems.

Sleep tracking data will be collected using consumer devices of the Charge series by Fitbit.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the feasibility of the planned study design and to evaluate the effect of Redormin® 500 on cognitive performance (reaction time, working memory) and psychological parameters with daily measures.

The primary objective of this study is to evaluate the feasibility of the study design to be able to design a confirmatory study.

The secondary objectives are to assess the influence of Redormin® 500 on cognitive performance (reaction time, working memory) and psychological parameters (subjective cognitive performance, stress levels, tiredness, mood, quality of life, and motivation; all of these measures with reference to the current day) with daily measures in the evening, and on sleep parameters and heart rate variability (HRV) as an objective measure for the stress level during day as assessed by the Fitbit tracker.

Safety objectives: Safety will be evaluated by obtaining and analysing adverse events during run-in period and treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male or female
* Age: 18-65 years old
* Occasional sleep problems (in average 1-2 nights per week, PSQI-score >5) with accompanying subjective cognitive problems (in average at least on one day per week) in the last month
* Fluent in German
* Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* DSM-V diagnosis of insomnia
* History of neurologic disorder
* Current psychiatric disorder
* Presence of moderately severe or severe depressive disorder (PHQ-9 ≥ 15)
* Current chronic intake of prescription drugs with psychotropic effects
* Current intake of OTC drugs for sleep or mood problems
* Presence of pain condition
* Diabetes mellitus
* Coronary Heart Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients completing the study | 21 days
  Percentage will be calculated by dividing the number of patients completing the study by number of patients interested in the advertisement

SECONDARY OUTCOMES:
Reaction time | each day for 21 days
  seconds
Subjective cognitive performance during the day (visual analogue scale) | each day for 21 days
  minimum value 1, maximum value 101, higher value means better cognitive performance
sleep duration | each day for 21 days
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Gerhards, Principal Investigator — University of Basel
Locations (1):
- Research Platform MCN University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schicktanz N, Gerhards C, Schlitt T, Aerni A, Muggler E, de Quervain D, Papassotiropoulos A, Boonen G, Drewe J, Butterweck V. Effects of a Valerian-Hops Extract Combination (Ze 91019) on Sleep Duration and Daytime Cognitive and Psychological Parameters in Occasional Insomnia: A Randomized Controlled Feasibility Trial. Brain Behav. 2025 Jun;15(6):e70600. doi: 10.1002/brb3.70600. PMID 40462685